CLINICAL TRIAL: NCT00740597
Title: Phase II Study of Preoperative Intensity-Modulated Radiation Therapy for Soft-Tissue Sarcomas
Brief Title: Intensity-Modulated Radiation Therapy in Treating Patients Undergoing Surgery for Stage IB, Stage II, or Stage III Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients were enrolled on the study
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07216; P30CA033572 (NIH); CHNMC-07216; CDR0000612344 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; adult alveolar soft-part sarcoma; adult epithelioid sarcoma; adult extraskeletal chondrosarcoma; adult extraskeletal osteosarcoma; adult fibrosarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult neurofibrosarcoma; adult rhabdomyosarcoma; dermatofibrosarcoma protuberans
MeSH Terms: conditions — Sarcoma; Sarcoma, Alveolar Soft Part; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Neurofibrosarcoma; Rhabdomyosarcoma; Dermatofibrosarcoma | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Blotting, Western; Neoadjuvant Therapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): pre-operative radiation + surgery PTV will receive a total dose of 50 Gy in 25 fractions, 2 Gy per fraction, 5 fractions per week, over approximately 5 weeks. Concurrently, the GTV2, if present, will receive 54 Gy in 25 fraction. Dose will be prescribed to the isodose volume that encompasses the PTV. All patients will be treated by 6 MV photon beam.
  Interventions: Genetic: gene expression analysis; Genetic: polymerase chain reaction; Genetic: western blotting; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: western blotting
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying the side effects of intensity-modulated radiation therapy and to see how well it works in treating patients undergoing surgery for stage IB, stage II, or stage III soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the wound complication rate in patients with stage IB-III soft tissue sarcoma (STS) treated with neoadjuvant intensity-modulated radiotherapy (IMRT).

Secondary

* Assess local control rate in patients treated with this regimen.
* Assess metastatic failure rate in patients treated with this regimen.
* Assess disease-free survival of patients treated with this regimen.
* Assess overall survival of patients treated with this regimen.
* Assess function and general health in these patients using the Musculoskeletal Tumor Society rating scale, Toronto Extremity Salvage Score, and the Short-Form 36.
* Determine changes in STS gene expression after IMRT by microarray analyses.
* Correlate, preliminarily, changes in STS gene expression with pathological and clinical outcomes.

OUTLINE: Patients undergo intensity-modulated radiotherapy (IMRT) once daily 5 days a week for 5 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery > 1 month after completion of IMRT.

Tumor tissue samples are collected at baseline and at the time of surgery for correlative laboratory studies. Samples are analyzed for gene expression by RNA microarray, real-time polymerase chain reaction, and western blotting.

After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma (STS) for which neoadjuvant or adjuvant radiotherapy is considered standard care

  * Stage IB-III disease
  * Primary or locally recurrent disease
* The following chemotherapy-sensitive STS histologies are excluded:

  * Primitive neuroectodermal tumor
  * Desmoplastic small round cell tumor
  * Synovial sarcoma
  * Myxoid round cell liposarcoma
  * Angiosarcoma
* No sarcomas for which surgical staging and adjuvant radiotherapy are considered standard care (e.g., uterine sarcomas, including leiomyosarcoma, malignant mixed Müllerian tumors, and endometrial stromal sarcoma)
* No retroperitoneal STS

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Able to complete the self-assessment questionnaires (may use translator service)
* Willing and able to undergo pre-treatment core needle biopsies
* Negative pregnancy test
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* Prior adjuvant chemotherapy for STS allowed provided patient has locally recurrent disease

  * At least 1 year since prior adjuvant chemotherapy
* No prior radiotherapy to the site of present STS
* No other concurrent cytotoxic chemotherapy, targeted therapy, or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D. Pezner, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 1
Completed | 0
Not Completed | 1
Not completed — insurance would not cover treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Wound Complication Rate
Description: Major wound complications up to 4 months post surgery include:
  Complications requiring a secondary operation under general or regional anesthesia for wound care.
  Seroma aspiration. Drain placement. Minor wound debridement and wound care. Readmission for wound care such as intravenous antibiotics. Persistent wound deep packing or wound vacuum assisted closure for greater than 120 days.
Time Frame: 1 year
Population: The one patient accrued to the study stopped treatment prior to completing treatment due to insurance denial.
Arm/Group | Arm 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Only one patients was on treatment for 5 days with no adverse events to report.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study closed 05/12/2010 (opened 7/25/2008): No patients were accrued and treated per protocol in nearly two years (2 patients were screened). The study was terminated by the IRB when the PI decided not to continue. Protocol objectives were not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes